CLINICAL TRIAL: NCT02373332
Title: Fatty Acid Regulation of Platelet Function in Diabetes
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Holinstat, Associate Professor of Pharmacology, University of Michigan
Other Study IDs: Michigan-114405A; R01HL114405 (NIH); ODS (Other: Office of Dietary Supplementation (NIH), co-funder)
Record Dates: First submitted 2015-02-20; First posted 2015-02-27 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Thrombosis; Type 2 Diabetes Mellitus
Keywords: platelets; 12-lipoxygenase; fatty acids; DGLA; DHA; EPA; 12-LOX
MeSH Terms: conditions — Thrombosis; Diabetes Mellitus, Type 2 | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Platelets, plasma, and whole blood will be assessed for platelet reactivity and thrombosis and stored for later analysis of protein expression. DNA will be stored for assessment of levels of gene products throught to play a role in platelet reactivity.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects for oxylipin effect Platelets from healthy donors will be assessed for regulation of platelet reactivity by fatty acids and 12-lipoxygenase oxylipins.
  Interventions: Other: omega-3 and -6 fatty acids and their 12-LOX oxylipins
- Type 2 diabetes mellitus (T2DM) patients: T2DM patients for oxylipin effect Platelets from healthy donors will be assessed for regulation of platelet reactivity by fatty acids and 12-lipoxygenase oxylipins.

INTERVENTIONS:
Other: omega-3 and -6 fatty acids and their 12-LOX oxylipins — platelets from healthy subjects and T2DM patients will be isolated from their blood and treated with omega-3 and -6 fatty acids and their 12-LOX oxylipins of those fatty acids followed by assessment of protection from agonist-induced platelet activation and thrombosis
  Groups: Healthy subjects

SUMMARY:
This study investigates the potential protective effects of altering fatty acid in the platelet as a method for prevention of platelet activation and thrombosis in type 2 diabetes mellitus. Fatty acids (omega-3 and omega-6) and their oxidized lipids will be evaluated for protection from agonist-mediated platelet activation in platelets from type 2 diabetics and healthy controls.

DETAILED DESCRIPTION:
12-lipoxygenase and essential fatty acids such as omega-3 and omega-6 have been shown to play important roles in regulating platelet activation, but the underlying mechanisms have not been fully elucidated as well as their true protection from thrombosis.

12-lipoxygenase inhibition prevents platelet activation in part by inhibiting 12-lipoxygenase oxidation of free fatty acids in the platelet. These oxidized fatty acids are known to play both a pro- and anti-thrombotic effect on platelets depending on the fatty acid. oxidation of arachidonic acid by 12-lipoxygenase results in a pro-thrombotic bioactive lipid whereas oxidation of the omega-6 fatty acid DGLA found in plant oil results in formation of a potent anti-thrombotic bioactive lipid. Determining the extent of protection from this and other bioactive lipids produced through 12-lipoxygenase will allow for a better understanding of which fatty acid supplementation may best protect from thrombosis.

Essential fatty acids such as omega-3 (DHA/EPA) and omega-6 (DGLA) appear to be protective. However the underlying mechanism for this potential protection is not well understood. Identifying the mechanism by which these supplements protect from platelet activation may identify new approaches to preventing thrombotic events in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects and T2DM patients
* African American and Caucasian
* T2DM patients on controlled medication (taking metformin)

Exclusion Criteria:

* Dietary supplement within 2 weeks of enrollment
* Fish and plant oil supplements 2 months prior to enrollment
* NSAIDS and aspirin 1 week prior to enrollment
* Smoking
* Cardiovascular event within 6 months prior to enrollment
* Other anti-platelet treatment including phosphodiesterase (PDE) and P2Y12R inhibitors
* Estimated Glomerular Filtration Rate (eGFR) below 30 (severe renal insufficiency)
* eGFR above 90

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 21-70. Both female and male and no preference for race or ethnicity. Subjects will abstain from anti-platelet therapy for 10 days. Health status will be confirmed by oral questioning and written questionnaire and confirmed following blood draw prior to evaluation of platelets with fatty acid or oxylipins.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
inhibition of platelet activation | one-time blood draw
  following blood draw, the ability of fatty acids or their oxylipins to inhibit platelet activation will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holinstat, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania